CLINICAL TRIAL: NCT00769990
Title: Phase I-II Trial of Genistein in Subjects Receiving Palliative External Beam Radiation Therapy for Osseous Metastases: A Study of Palliation of Symptoms and Quality of Life
Brief Title: Genistein in Treating Patients Undergoing External-Beam Radiation Therapy for Bone Metastases
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No patient accrual.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008LS035; UMN-0803M29541 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2011-07

CONDITIONS: Breast Cancer; Kidney Cancer; Lung Cancer; Melanoma; Metastatic Cancer; Pain; Prostate Cancer
Keywords: bone metastases; pain; recurrent breast cancer; stage IV breast cancer; recurrent prostate cancer; stage IV prostate cancer; recurrent melanoma; stage IV melanoma; recurrent renal cell cancer; stage IV renal cell cancer; recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Breast Neoplasms; Kidney Neoplasms; Lung Neoplasms; Melanoma; Neoplasm Metastasis; Pain; Prostatic Neoplasms; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Genistein; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Genistein (Experimental): Patients treated with Genistein who are going to undergo palliative radiation treatments for painful boney metastases.
  Interventions: Dietary Supplement: genistein; Radiation: radiation therapy

INTERVENTIONS:
Dietary Supplement: genistein — Genistein will be taken orally once daily as 500 mg capsules throughout the study (60 days).
  Other Names: Bonistein
Radiation: radiation therapy — A course of palliative external beam radiation therapy -performed within 8 weeks prior to start of the study.

SUMMARY:
RATIONALE: Genistein may increase the effectiveness of radiation therapy in treating pain caused by bone metastases.

PURPOSE: This phase I/II trial is studying the side effects of genistein and to see how well it works in treating patients undergoing external-beam radiation therapy for pain caused by bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether genistein is safe when administered in combination with palliative external beam radiotherapy in patients with osseous metastases.
* To determine the time to pain relief, duration of pain relief, and degree of pain relief in patients treated with this regimen.
* To determine the incidence of pathologic fractures in patients treated with this regimen.
* To determine the effect of this regimen on quality of life measures in these patients.

OUTLINE: This is a multicenter study.

Patients undergo external beam radiotherapy once daily on days 1-10. Patients also receive oral genistein once daily on days 1-60.

Patients complete pain and quality-of-life questionnaires periodically.

After completion of study therapy, patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant solid tumor, including any of the following:

  * Breast cancer
  * Lung cancer
  * Kidney cancer
  * Melanoma
  * Prostate cancer
* Radiographic evidence* of bone metastasis within the past 8 weeks NOTE: *Acceptable studies include plain radiograph, radionuclide bone scan, CT scan, and MRI
* Has pain that appears to be related to the radiographically documented metastasis, in the opinion of the treating physician, AND a decision has been made by the responsible clinician that a course of palliative external beam radiotherapy is appropriate treatment

  * "Worst pain score" of > 5 on a scale of 10 as scored on the pain assessment questionnaire (BPI) (question #3: 0 = no pain; 10 = worst possible pain) OR taking narcotic medications with an oral morphine equivalent dose of > 60 mg/day
  * No painful metastases to the skull, hands, or feet
* Eligible treatment sites include any of following:

  * Weight-bearing sites:

    * Pelvis (excluding pubis)
    * Femur
    * Sacrum and/or sacroiliac joints
    * Tibia
  * Non-weight-bearing sites:

    * Up to 5 consecutive cervical, thoracic, or lumbar vertebral bodies
    * Lumbosacral spine
    * Up to 3 consecutive ribs
    * Humerus
    * Fibula
    * Radius ± ulna
    * Clavicle
    * Sternum
    * Scapula
    * Pubis
* If multiple osseous sites are treated, the treatment site is included as weight-bearing if any of the sites include the pelvis, sacrum, femur, or tibia

  * Treatment of multiple osseous sites allowed only if those sites can be included in ≤ 3 treatment sites
* Patients with painful metastases that are contiguous but do not fit into the definition of a site listed above are eligible but are considered to have 2 treatment sites
* No vertebral metastases with clinical or radiographic evidence of spinal cord or cauda equina compression/effacement
* No primary hematologic malignancies (e.g., lymphoma)
* Hormone receptor status (for patients with breast cancer):

  * Estrogen receptor-negative tumor
* Menopausal status not specified
* Karnofsky performance status 40-100%
* Life expectancy ≥ 3 months
* ALT normal
* Bilirubin normal
* Serum creatinine normal (≤ 1.8 mg/dL for males and ≤ 1.5 mg/dL for females)
* Free T4 and thyroid-stimulating hormone normal
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pathologic fracture or impending fracture of the treatment site
* No history of primary hyperparathyroidism
* No malabsorptive disease or chronic diarrhea
* No history of sarcoidosis or tuberculosis

Exclusion Criteria:

* Less than 30 days since prior systemic radioisotopes for pain, including Strontium-90 (^90Sr) or Samarium (^153Sm)
* Less than 30 days since prior antibiotics
* Less than 30 days since prior initiation of systemic therapy (e.g., hormonal therapy, chemotherapy, or immunotherapy)
* Less than 90 days since prior intravenous bisphosphonate therapy

  * Concurrent oral bisphosphonates allowed
* Prior radiotherapy or palliative surgery to the painful sites
* Concurrent surgical fixation of the bone
* Concurrent treatment to the skull, hands, or feet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety | At completion of first 6 patients
  Frequency of severe (grade 3) toxicities

SECONDARY OUTCOMES:
Time to pain relief, duration of pain relief, and degree of pain relief
Incidence of pathologic fractures
Effect of treatment on quality of life measures as assessed by the BPI and FACT-G

CONTACTS AND LOCATIONS:
Overall Officials: Shalamar Sibley, MD, MPH, Principal Investigator — Masonic Cancer Center, University of Minnesota